CLINICAL TRIAL: NCT00003870
Title: Radiolabeled BC8 (Anti-CD45) Antibody Combined With Cyclophosphamide and Total Body Irradiation Followed by HLA-matched Related or Unrelated Stem Cell Transplantation as Treatment for Advanced Acute Lymphocytic Leukemia
Brief Title: Monoclonal Antibody Therapy, Cyclophosphamide, and Total-Body Irradiation Followed by Peripheral Stem Cell Transplantation in Treating Patients With Advanced Recurrent Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1298.00; FHCRC-1298.00; NCI-H99-0029; CDR0000067034 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Methotrexate; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Radiation: iodine I 131 monoclonal antibody BC8
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy, cyclophosphamide, and total-body irradiation followed by peripheral stem cell transplantation in treating patients who have advanced recurrent acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy and toxicity of iodine I 131 monoclonal antibody BC8, cyclophosphamide, and total body irradiation in patients with advanced acute lymphocytic leukemia who are receiving HLA matched related or unrelated bone marrow transplantation. II. Determine the maximum tolerated dose (MTD) of iodine I 131 monoclonal antibody BC8 in these patients. III. Estimate the MTD of radiation delivered by iodine I 131 monoclonal antibody BC8 to the marrow. IV. Study the influence of marrow cellularity, level of antigen expression by leukemic cells, and degree of antigen saturation by antibody on the biodistribution of iodine I 131 monoclonal antibody BC8 in these patients.

OUTLINE: This is a dose-escalation study. All patients receive a test dose of iodine I 131 monoclonal antibody BC8 (MOAB BC8) IV over several hours 6-14 days prior to the therapeutic dose. Patients receive the therapeutic dose of iodine I 131 MOAB BC8 IV over several hours on day -11, total body irradiation over 30-40 minutes twice a day on days -6 to -4, and cyclophosphamide IV over 1 hour on days -3 and -2. Patients undergo allogenic bone marrow transplantation on day 0. Patients receive intrathecal methotrexate twice prior to transplantation and then every other week for 4 weeks beginning on day 32 posttransplant. Cohorts of 4 patients receive escalating doses of iodine I 131 monoclonal antibody until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 4 patients experience dose-limiting toxicity. Patients are followed for the first 100 days, at 6, 9 and 12 months, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed acute lymphocytic leukemia that is beyond first remission or is refractory Relapsed disease must be CD45 positive Patients in remission may be CD45 negative

PATIENT CHARACTERISTICS: Age: 2 to 55 Performance status: Not specified Life expectancy: More than 60 days Hematopoietic: Circulating blast count less than 10,000/mm3 (control with hydroxyurea or similar agent allowed) Hepatic: Bilirubin less than 1.5 mg/dL AST less than 1.5 times upper limit of normal (ULN) Must have no veno-occlusive liver disease Renal: Creatinine less than 2.0 mg/dL OR less than 1.5 times ULN for age Other: No active infection HIV negative No circulating antimouse immunoglobulin antibodies Must be able to tolerate diagnostic or therapeutic procedures (e.g., radiation isolation)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to maximum tolerated levels to any normal organ Surgery: Not specified

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-02; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Christine Matthews, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington